CLINICAL TRIAL: NCT05150054
Title: Magnetocardiography as a Noninvasive Diagnostic Strategy for Suspected Coronary Microvascular Dysfunction
Brief Title: MCG as a Noninvasive Diagnostic Strategy for Suspected Coronary Microvascular Dysfunction
Acronym: MICRO
Status: Completed | Type: Observational
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1000-6
Record Dates: First submitted 2021-11-18; First posted 2021-12-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Coronary Microvascular Dysfunction; Ischemic Non-Obstructive Coronary Artery Disease
Keywords: INOCA; Magnetocardiography; CardioFlux; MCG; Coronary Microvascular Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CardioFlux — Not an intervention

SUMMARY:
According to the Women's Ischemic Syndrome Evaluation database, there are approximately 3 to 4 million women and men who present with signs and symptoms that are suggestive of myocardial ischemia, however they have no obstructive coronary artery disease (INOCA). INOCA is defined as patients presenting with signs or symptoms of ischemia but no obstructive artery disease. Women are more likely than men to die from cardiovascular disease and more likely to present with no obstructive coronary artery disease. Patients who present with signs and symptoms suggestive of INOCA/MINOCA are also presenting with Coronary Microvascular Dysfunction (CMD). Coronary Microvascular Dysfunction is a dysfunction in the epicardial and/or microvascular endothelial and/or nonendothelial that limits myocardial perfusion. Today, there is no routinely offered/available noninvasive test that is used for the diagnosis of CMD, significantly hindering the ability to identify the disease in the standard of care. Magenetocardiography (MCG) has the opportunity to use its noninvasive imaging techniques to provide early management of CMD. Magnetocardiography (MCG) is a noninvasive imaging modality that has been extensively studied, over the past several decades, as a diagnostic imaging solution for various forms of cardiovascular disease. MCG measures the magnetic field that arises from the electrical activity of the heart's pacemaker activity, the very same activity which yield surface electric field potentials as measured by the electrocardiogram. Since MCG is a functional assessor of repolarization heterogeneity, it is hypothesized that MCG may be a useful frontline diagnostic to identify CMD in patients who would otherwise have normal coronary CT angiograms and/or stress tests. The proposed study intends to study the diagnostic accuracy of MCG in this population, with the goal of providing early and noninvasive insights for management of CMD. There will be a 12-month duration of the study where the investigators propose to collect MCG scans from approximately 150 patients who present to the Genetesis facility for a 15-minute CardioFlux scan appointment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment
2. Signs and symptoms of chest pain that prompted further evaluation by either a heart angiogram or a scan of the heart (coronary CT angiogram) within the previous 5 years
3. Willing to provide written informed consent
4. Non-obstructive CAD defined as 0 to 49% diameter reduction of a major epicardial vessel or a FFR>0.80
5. Scheduled for CRT
6. No cardiac medications in the last 24 hours of an MCG-CF scan (with the exception of the patients enrolled in the data development set)

Exclusion Criteria:

1. Patients unable to fit into device
2. Non-ambulatory patients
3. Patients who meet device contraindications
4. Patients unable to lie supine for 5 minutes
5. History of noncompliance (with medical therapy, protocol, or follow-up)
6. History of non-ischemic dilated or hypertrophic cardiomyopathy
7. Documented acute coronary syndrome (ACS) within previous 30 days
8. Left ventricular ejection fraction (LVEF) <40%, New York Heart Association heart failure (NYHA HF) class III-IV, or hospitalization for Reduced ejection fraction (HFrEF) within 180 days
9. Stroke within previous 180 days or intracranial hemorrhage at any time
10. End-stage renal disease, on dialysis, or estimated glomerular filtration rate (eGFR) <30 ml/min.
11. Severe valvular disease or likely to require surgery/Transcatheter aortic valve replacement (TVAR) within 3 years
12. Life expectancy <3-yrs. due to non-cardiovascular comorbidity
13. Enrolled in a competing clinical trial
14. Prior intolerance to both an ACE-I and ARB
15. If intolerant to a statin unless taking a PCSK9 as a statin replacement by their clinical provider
16. Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting with signs and symptoms of chest pain that prompted further evaluation by either a heart angiogram or a scan of the heart (coronary CT angiogram) within the previous 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CardioFlux | 12 months
  Analyzing the diagnostic accuracy of CardioFlux in determining the presence of coronary microvascular dysfunction

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Ascension St. John, Detroit, Michigan
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Genetesis Facility, Mason, Ohio

IPD SHARING:
Plan to Share IPD: No